CLINICAL TRIAL: NCT04245384
Title: Dietitian Online - Internet-based Dietetic Treatment Within Health Care Services
Acronym: DiOn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Umeå University (Other)
Collaborators: Västerbotten County Council, Sweden (Other Government); Forte (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UmUDiOn
Record Dates: First submitted 2020-01-21; First posted 2020-01-28 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Overweight and Obesity
Keywords: dietetics; telemedicine; dietitian
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based treatment (Experimental): Internet-based dietetic treatment with video calls, no physical meetings
  Interventions: Other: Internet-based dietetic treatment with video calls
- Standard treatment (Active Comparator): Dietetic treatment with physical meetings
  Interventions: Other: Traditional dietetic treatment

INTERVENTIONS:
Other: Internet-based dietetic treatment with video calls — The dietitian meets the patient through video calls, no physical meetings
  Arms: Internet-based treatment
Other: Traditional dietetic treatment — The dietitian meets the patient through physical meetings
  Arms: Standard treatment

SUMMARY:
The project aims to investigate the effect of internet-based dietetic treatment (IDT) on patients, dietitians, and society.

The project will show:

* If IDT is equivalent to traditional dietetic treatment with physical meetings
* Patients' attitudes to, and experiences of, meeting a dietician through video calls
* How the dietician's work environment and working methods are affected by IDT
* If there are subgroups of patients where IDT is more or less appropriate
* Health economic and environmental consequences of IDT The major shortage of dietitians leaves patients with non-communicable diseases (NCD) without qualified dietary treatment. In a pilot study, the investigators have shown that IDT has great potential to streamline healthcare and increase accessibility. In the project Dietitian online, the investigators will conduct an RCT with 400 NCD-patients allocated to either IDT or standard dietetic treatment to see if IDT affect treatment outcome and whether IDT is appropriate for everyone. Even though internet-based treatment (IT) increases rapidly in society, there is little knowledge about the patients' experiences and how healthcare personnel incorporates IT in their daily work. The investigators will conduct qualitative studies to meet this knowledge gap. General assumptions are that IT is beneficial for society, both economically and environmentally, but very few studies have been done. The project will incorporate a full health-economic evaluation, including environmental impact.

ELIGIBILITY:
Inclusion Criteria:

* seeking/being referred to a dietitian for the treatment of obesity (BMI≥25) or obesity in combination with:

  * type 2 diabetes (HbA1c>48mmol/mol) and/or
  * elevated blood lipids (total cholesterol >4,5 mmol/l and/or LDL >2,5 mmol/l and/or triglycerides >2,0 mmol/l) and/or
  * high blood pressure (>140/90 hg)

Exclusion Criteria:

* other diagnoses requiring/might require nutritional treatment (eg cancer, COPD)
* dementia
* severe impairment of sight, hearing, or other disability where internet-based dietetic treatment is deemed difficult
* pregnancy
* need for interpreter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in dietary intake | Change from baseline to three, six and twelve months after first treatment session
  Dietary intake will be assessed using the Swedish National Food Administrations Food Index (minimum value 0, maximum value 12, higher score indicates a healthier diet). Intake of fruit and vegetables in grams, as well as intake of discretionary calories (sweets, snacks, fast food, sugary drinks, pastries), will also be assessed.

SECONDARY OUTCOMES:
Change in participant alliance to dietitian | Change from baseline to three and six months after first treatment session
  Alliance between patient and dietitian, measured with Working Alliance Inventory - Short (WAI-S, minimum value 12, maximum value 84, higher score indicates higher alliance to dietitian)
Change in participant activation | Change from baseline to six months after first treatment session
  Patient activation (readiness to behavioral change), measured with Patient Activation Measure (PAM, (minimum value 0, maximum value 100, higher score indicates a higher activation (better)).
Change in participant motivation | Change from baseline to three. six and twelve months after first treatment session
  Patient motivation (personal motivation to behavioral change), measured with VAS-scale 0-100, where higher score indicates higher motivation to behavioral change.

OTHER OUTCOMES:
Change in body weight | Change from baseline to three, six and twelve months after first treatment session
  Self reported body weight
Change in physical activity | Change from baseline to three, six and twelve months after first treatment session
  Physical activity, measured as average physical activity level (PAL) at work and at leisure time using a validated two-question questionnaire. PAL-levels from the questionnaire range between 1.4 - 2.3, where a higher score indicates higher physical activity
Change in health-related quality of life | Change from baseline to six months after first treatment session
  Health-related quality of life, measured with EQ-5D (minimum value 0, maximum value 1 where a higher value indicates higher quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Petra M Rydén, PhD, Principal Investigator — Umea university

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Official website for the project (only in Swedish) — http://www.umu.se/dion